CLINICAL TRIAL: NCT03304080
Title: A Multicenter, Phase I/II Trial of Anastrozole, Palbociclib, Trastuzumab and Pertuzumab in HR-positive, HER2-positive Metastatic Breast Cancer
Brief Title: Anastrozole, Palbociclib, Trastuzumab and Pertuzumab in HR-positive, HER2-positive Metastatic Breast
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Herbert Irving Comprehensive Cancer Center (Other); Weill Medical College of Cornell University (Other); NYU Langone Health (Other)
Responsible Party: Principal Investigator, Amy Tiersten, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0919
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: Breast Neoplasms; Breast Diseases; Palbociclib; Trastuzumab; Pertuzumab; Hormone Antagonists; Anastrozole; Arimidex; Ibrance; Perjeta
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Anastrozole; palbociclib; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HR-positive, Her2-positive Metastatic Breast Cancer (Experimental): Women and men with HR-positive, HER2-positive Metastatic Breast Cancer on trial of anastrozole, palbociclib, trastuzumab and pertuzumab
  Interventions: Drug: Anastrozole; Drug: Palbociclib; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Anastrozole — 1 mg orally daily, day 1 to day 28
  Other Names: Arimidex
Drug: Palbociclib — Dose I: 100 mg orally daily, day 1 to day 21, then 7 days off in a 28 day cycle (Phase 1 only) Dose II: 125 mg orally daily, day 1 to day 21, then 7 days off in a 28 day cycle
  Other Names: Ibrance
Drug: Trastuzumab — 8 mg/kg IV initial loading dose, followed by 6 mg/kg IV every 21 days
  Other Names: Herceptin
Drug: Pertuzumab — 840 mg IV followed by a maintenance dose of 420 mg IV every 21 days
  Other Names: Perjeta

SUMMARY:
This is a multicenter, phase I/II trial of anastrozole, palbociclib, trastuzumab, and pertuzumab is proposed as first-line therapy in metastatic hormone receptor-positive, HER2-positive breast cancer patients. In this phase I/II clinical trial, the researchers aim to establish the safety and efficacy of dual HER2 therapy in combination with palbociclib and anastrozole, which represents a novel and all biologic approach to the treatment of HR+, HER2+ metastatic breast cancer. Additionally, the researchers aim to examine potential biomarkers of response to palbociclib including cyclin D1, cyclin E1 and cyclin E2 expression levels, CDK 2, 4, and 6 levels, phosphorylated retinoblastoma expression and p16 levels. The researchers intend to use RNA sequencing to assess for other predictors of response in an unbiased manner to see if this correlates with inhibition of Ki-67 and phosphorylated retinoblastoma expression as well as evaluate for potential mechanisms of resistance.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with metastatic breast cancer, measurable or evaluable disease including bone metastasis only (as per the Response Evaluation Criteria in Solid Tumors [RECIST] v1.1)
* No prior systemic treatment for metastatic breast cancer
* Pathologic confirmation of metastatic breast cancer diagnosed by core needle biopsy
* Metastatic breast cancer with any evidence of ER or PR positivity in ≥ 1% cells in biopsy specimens from either a primary or metastatic site
* Evidence of HER2 positive metastatic breast cancer in either a primary or metastatic site, if 3+ by an IHC method defined as uniform membrane staining for HER2 in 10% or more of tumor cells or demonstrate HER2 gene amplification by an ISH method (single probe, average HER2 copy number ≥6.0 signals/cell; dual probe HER2/CEP17 ratio ≥2.0 with an average HER2 copy number ≥4.0 signals/cell; dual probe HER2/chromosome enumeration probe (CEP) 17 ratio ≥2.0 with an average HER2 cop number <4.0 signals/cell; and HER2/CEP17 ratio <2.0 with an average HER2 copy number ≥6.0 signals/cell) or amplified by FISH > 2.0. High average copy number of HER2 (≥6.0 signals/cell) is considered positive regardless of the HER2/CEP17 ratio.
* Women or men 18 years and older
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Stable brain metastasis allowed (>2 weeks, clinically stable post treatment with surgery +/- radiation or radiation alone and off steroids)
* Transthoracic echocardiogram with ejection fraction > 50%
* Postmenopausal status or receiving ovarian ablation with a GnRH agonist such as goserelin or leuprolide. Postmenopausal status is defined by any one of the following criteria:

  * Prior bilateral oophorectomy.
  * Prior ovarian radiation for the purpose of ablation.
  * Age ≥ 60 years.
  * Age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, or ovarian suppression) and FSH, LH, and estradiol in the postmenopausal range per local normal.
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* A baseline CT chest/abdomen/pelvis and bone scan or PET/CT
* Negative serum or urine pregnancy test within 7 days prior to starting treatment
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Note: Recommended methods of birth control are: The consistent use of an intrauterine device (IUD), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), sexual abstinence (no sexual intercourse) or sterilization.

Men must agree to use a condom and not father a child for the duration of the study and for 90 days after completion of therapy

Laboratory values (≤ 28 days prior to registration)

* Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
* Platelet Count ≥ 75,000/ mm3
* Hg >9 g/dL
* Total Bilirubin ≤1.5 x upper limits of normal (ULN)
* Serum ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN in patients with liver metastasis)
* Creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* HER2 negative metastatic breast carcinoma defined as 0 or 1+ by IHC or with a FISH ratio (HER2 gene copy/ chromosome 17) <2 if IHC 2+ by local institution standard protocol
* Any prior treatment for metastatic breast cancer. (excluding radiation therapy for the purpose of ovarian ablation). Note: Prior adjuvant therapy with trastuzumab and pertuzumab is permitted after a 6 month window following completion of adjuvant therapy has passed.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks of the start of study drug (including chemotherapy, radiation therapy, and biologics). Patients who have received prior endocrine therapy for fertility purposes will be eligible.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 2 weeks
* Co-administration with strong CYP3A4 inducers (e.g., phenytoin, rifampin, carbamazepine, St John's Wort, bosentan, efavirenz, etravirine, modafinil, and nafcillin), strong CYP3A4 inhibitors (e.g., clarithromycin, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, and voriconazole), and CYP3A4 substrates (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, everolimus, fentanyl, pimozide, quinidine, sirolimus and tacrolimus). For a current table of Substrates, Inhibitors and Inducers please access the following website:http://www.fda.gov/Drugs/DevelopmentApprovalProcess/" See Appendix C.
* Uncontrolled brain metastases
* Leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 89% or less at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of palbociclib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Ongoing alcohol or drug addiction
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to starting treatment)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib, anastrozole, trastuzumab or pertuzumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | up to 3 months
  The dose-limiting toxicity (DLT) for palbociclib when administered in combination with anastrozole, trastuzumab and pertuzumab. A DLT will be defined as:
  * Grade 3 or 4 non-hematologic toxicity
  * Grade 3 neutropenia lasting greater than 21 days
  * Grade 3 or 4 neutropenia with neutropenic fever or
  * Grade 4 hematologic toxicity events experienced within the first 4 weeks (1 cycle) of study treatment. These will be assessed via the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI's CTCAE) v4.0 toxicity criteria.
Maximum Tolerated Dose (MTD) | up to 3 months
  The maximum tolerated dose (MTD) for palbociclib when administered in combination with anastrozole, trastuzumab and pertuzumab. If > 33 % of patients experience a dose limiting toxicity (DLT) at any dose level, the dose level below that level will be considered the MTD. Or if the highest level has been reached and ≤ 33% of patients have experienced dose limiting toxicity (DLT), that will be considered the MTD.
Clinical Benefit Rate (CBR) | average of 6 months
  CBR will be measured by the percentage of patients whose cancer shrinks or remains stable over the duration of the study. This will be measured as the sum of complete response, partial response, and stable disease for greater than or equal to 6 months.

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  The time from the start of treatment until confirmed disease progression or death from any cause, whichever occurs first.
Incidence of adverse events | 2 years
  incidence of adverse events as graded by the NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Mount Sinai Beth Israel Comprehensive Cancer Center West, New York, New York
  - Perlmutter Cancer Center NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - New York Presbyterian Columbia Irving Comprehensive Cancer Center, New York, New York
  - New York Presbyterian Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Data collected during the course of this clinical trial will primarily be shared with other investigators and University staff, the IRB, FDA, and other reporting agencies, and/or transferred to other collaborators. Prior to transfer, the data collected must comply with, and must be limited by, the MSH's guidelines for Protecting the Rights and Privacy of Human Subjects.